CLINICAL TRIAL: NCT06637124
Title: Blood Flow Restriction with Different Loads Versus Moderate Resistive Exercises in Patients with Knee Osteoarthritis: a Double Blinded Randomized Controlled Trial
Brief Title: Different Levels of Blood Flow Restriction Versus Moderate Intensity Exercises in Patients with Knee Osteoarthritis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Farah Fouad Gomaa El Gamal, Masters Degree Student in Faculty of Physical Therapy, Cairo University, Cairo University
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P.T.REC/012/005029
Record Dates: First submitted 2024-09-24; First posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-01

CONDITIONS: Knee Osteoarthritis; Blood Flow Restriction Therapy
Keywords: Blood Flow Restriction; Knee osteoarthritis; Moderate Intenstity Exercise
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- 50% Blood Flow Restriction Group (Experimental): The Blood Flow Restriction device will be set to restrict blood flow at level of 50% of arterial occlusion pressure at rest.
  Blood Flow Restriction sessions will be 5 sets of 5 mins of occlusion and 3 mins of free flow , 2 sessions per week for eight weeks exercises to assess its effects on knee osteoarthritis-related outcomes.
  Interventions: Device: Blood Flow Restriction Therapy Device
- 70% Blood Flow Restriction Group (Experimental): The Blood Flow Restriction device will be set to restrict blood flow at level of 70% of arterial occlusion pressure at rest.
  Blood Flow Restriction sessions will be 5 sets of 5 mins of occlusion and 3 mins of free flow , 2 sessions per week for eight weeks exercises to assess its effects on knee osteoarthritis-related outcomes.
  Interventions: Device: Blood Flow Restriction Therapy Device
- Moderate Intensity Exercise training Group (Active Comparator): Patients assigned to this group will receive strengthening of the lower limb musculature through moderate intensity resistance training (60% of 1RM) for a total of 16 treatment sessions according to exercise guidelines for seniors with OA.
  MIRT protocols consists of 3 sets for every exercise, 12 repetitions per set, rest period between sets 2 mins, 2 session per week for 8 weeks.
  Resistance exercises will be performed using a 45° leg-press machine, 90°-0° of knee flexion knee extension machine, leg curl machine and calf raise machine.
  Interventions: Device: 45° leg-press machine, 90°-0° of knee flexion knee extension machine, leg curl machine and calf raise machine.

INTERVENTIONS:
Device: Blood Flow Restriction Therapy Device — Blood Flow Restriction (BFR) therapy involves units use standardized cuffs of varying widths and lengths which are physically attached to the devices and provide the capability of precisely controlling the amount of pressure applied to each limb during exercise or at rest.
  We will be using Smart Cuffs® 4.0 which allows for a fast, hassle-free personalized pressure calculation. With the built-in pressure sensor and on-board computer, it will calculate and set the optimal pressure for each participant's limb. There is no need for an external doppler probe or hand pump. Made in the USA, SmartCuffs® are registered with the FDA as a Class 1 Medical Device.
  Blood flow restriction therapy is commonly paired with resistive training, so this study will explore the effect of blood flow restriction at rest for patients with osteoarthritis at different restriction levels (50% for first group and 70% for second group).
  Other Names: Smart cuffs 4.0
  Arms: 50% Blood Flow Restriction Group; 70% Blood Flow Restriction Group
Device: 45° leg-press machine, 90°-0° of knee flexion knee extension machine, leg curl machine and calf raise machine. — Patients assigned to group will receive strengthening of the lower limb musculature through moderate intensity resistance training (60% of 1RM) using a 45° leg-press machine, 90°-0° of knee flexion knee extension machine, leg curl machine and calf raise machine.
  Arms: Moderate Intensity Exercise training Group

SUMMARY:
This clinical trail will be conducted to investigate the effect of blood flow restriction (BFR) with different load levels between low blood occlusion percentage (50%) group and high blood occlusion percentage (70%) compared to moderate intensity training (60% of 1 RM) in patients with chronic knee osteoarthritis.

The main questions it aims to answer are:

1. Will there be no difference between the effect of (70% vs 50%) of BFR versus traditional moderate resistive training exercises on pain intensity in knee osteoarthritis ?
2. Will there be no difference between the effect of (70% vs 50%) of BFR versus traditional moderate resistive training exercises on quadriceps muscle strength in knee osteoarthritis ?
3. Will there be no difference difference between the effect of (70% vs 50%) of BFR versus traditional moderate resistive training exercises on rate of perceived exertion in knee osteoarthritis ?
4. Will there be no difference between the effect of (70% vs 50%) of BFR versus traditional moderate resistive training exercises on functional ability in knee osteoarthritis ?
5. Will there be no difference between the effect of (70% vs 50%) of BFR versus traditional moderate resistive training exercises on physical function in knee osteoarthritis ?

All participants will receive:

1. 16 sessions of supervised intervention 2 times per week for 8 weeks.
2. The assessment will be at 3 time points, baseline and at 4 weeks and at 8 weeks.

DETAILED DESCRIPTION:
Knee osteoarthritis (KOA) is a prevalent degenerative musculoskeletal condition that primarily causing pain, stiffness, and disability. It is a multifactorial disease influenced by a combination of genetic, biomechanical, and environmental factors Osteoarthritis Research Society International (ORSI) recommended strength training as a possible treatment method to slow progression of knee OA. Strength training, as recommended by the American College of Sports Medicine (ACSM), must be performed at a minimum resistance training load of 60% to 70% 1-repetition maximum (1RM) for strength improvement.

Only 13% of older patients with knee OA satisfactorily can perform moderate to vigorous physical activity.

Unfortunately, risk factors of knee OA (as obesity, knee pain, knee injury/surgery) also contribute to a perceived reduced tolerance to the resistive training programs recommended for eliciting strength gains.

An alternative to traditional strength training that may be well tolerated by patients with Knee OA is Blood flow restriction (BFR) training.

This reduced blood flow creates a unique physiological environment, inducing a state of metabolic stress and cellular hypoxia in the muscles.

Although the advantages of BFRT in musculoskeletal rehabilitation that reported in the literature, there are conflicting results compared to traditional exercises, as the different protocols parameters, exercises, high risk of bias across previous studies contribute to different conclusions.

Consequently, it raises the question if BFR without exercises can be effective in comparison with traditional exercises that focus on having an efficient intensity to produce muscle strength gain.

Yet, up to authors knowledge, no study has assessed whether BFR at rest could also promote similar gains in muscle strength for the knee OA treatment, which theoretically would increase patient's adherence to KOA treatment based on conclusions of systemic review of BFR without exercises for immobilized patients after orthopedic surgery (Cerqueira et al., 2019).

Another relevant issue is the proper blood flow restriction level for optimal results. Thus, pushes the need for determining a pressure load with the least adverse effects.

Therefore, the main purpose of this study is to assess different protocols of BFR without additional exercises compared to MI-RT for pain reduction in patients with KOA. The secondary purpose is to compare two load levels (70% vs 50%) of BFRT regarding pain, quadriceps muscle strength, rate of perceived exertion, self reported physical function, and functional ability.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with chronic knee osteoarthritis referred by orthopedic surgeons participants of both genders age are 40-65.
* Patients with grade 2 and 3 OA of the knee, according to radiologic evaluation
* If both knees diagnosed as OA, the most affected one will be selected.
* Diagnosis of Knee OA who had knee pain and functional disabilities for at least three months, according to American College of Rheumatology classification at screening visit.
* Visual Analogue Scale (VAS) at rest score of ≥40 mm.
* Arabic version of the western WOMAC (ArWOMAC) scores (average 37).
* Moderate Physical activity score on the IPAQ (between 3.0 and 7.9 METS).

Exclusion Criteria:

* Moderate to significant knee synovitis
* Hot or red knee
* History and/or physical examination findings compatible with the internal derangement of knee.
* Knee pain that is initiated or increased with knee activity/exercise and finished or decreased with knee resting.
* Other muscular, articular, or neurological condition affecting lower limb function.
* Patients with any previous knee surgeries or fractures of lower limb
* Patients who had undergone arthroscopy or treatment with intra-articular hyaluronic acid during the previous 6 months.
* Psychological or psychiatric disorders that may affect a subject's participation in the study.
* Participants with congenital musculoskeletal lower limb deformity.
* Participated in other intervention studies on the past 6 months to screening
* Participants with contraindications to blood flow Restriction Training.

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2024-07-15 (Actual); Primary Completion 2024-10-06 (Estimated); Study Completion 2024-10-30 (Estimated)

PRIMARY OUTCOMES:
Change in pain intensity | Measured 3 times at basline, 4 weeks and 8 weeks
  Measured by the Visual Analog Scale (VAS)which is a pain intensity assessment tool.
  * Represented with a 10 cm line with 0 indicating no pain and on the other end 10 indicating severe pain.
  * The patient is asked to move a marker on the line to the position which best describes their pain.
  * That it will serve as a subjective measure of their current level of knee pain intensity.
  The closer the mark to zero is better.
Measure change in quadriceps muscle strength | Measured 3 times at baseline, 4 weeks and 8 weeks
  Hand-held dynamometer (HHD) will be used to measure the strength in quadriceps muscle.
  * The maximum force or pressure exerted by the quadriceps muscle during the contraction will be recorded.
  * Typically, this measurement is expressed in kilograms (kg) and then transferred to Newtons (N)
  * To enhance reliability, 3 trials may be conducted, and average will be taken to obtain a more representative measurement of muscle strength.
  * The higher the measurement the higher the muscle strength.

SECONDARY OUTCOMES:
Change in functional ability | Measured 3 times at baseline, 4 weeks and 8 weeks
  Measured by Timed Up and Go Test (TUG) to assess participants' mobility, balance, and functional performance.
  * The time taken by the patient to complete the entire sequence from rising from the chair to returning to a seated position will be measured.
  * This time will be recorded in seconds, representing the TUG test score.
  * 3 times will be conducted to ensure the accuracy of the TUG test score.
  * The average time from these trials will be calculated for a more reliable result.
  * High Risk of fall (>13.5 seconds)
  * None/low/moderate (<13.5 seconds) The lower the number the better as it represents better mobility, balance and functional performance.
Change in physical function levels | Measured 3 times at baseline, 4 weeks and 8 weeks
  Measured by Arabic version of Western Ontario McMaster Universities Osteoarthritis Index for Knee Function (ArWOMAC).
  The WOMAC questionnaire will be handed out to the participants. They will be informed that it consists of a series of questions related to their knee symptoms and how these symptoms affect their daily activities.
  WOMAC is assigned a numerical score of 0-4 corresponding to severity (none, mild, moderate, severe, and extreme). The minimum score is 0, and the maximum score is 96 (20 points for pain, 8 points for joint stiffness, and 68 points for physical function).
  The lower the score the better.
Change in Rate of perceived exertion scale (RPE) | Measured 3 times at basline , 4 weeks and 8 weeks
  Measured by Arabic version of Omnibus Resistance Exercise 0-10 (OMNI-RES) as a scale for measuring an individual's effort and exertion, breathlessness and fatigue during physical work.
  * The OMNI Picture System is a collection of category scales used for rating of perceived exertion (RPE) as the subjective intensity of a person's feelings of effort, strain, discomfort, and/or fatigue when engaged in exercise or other physical activities.
  * With OMNI exertion scales, users select a number from 0 to 10 that best corresponds to their perceived intensity of physical exertion.
  * 0 represents extremely easy and 10 represents extremely hard.
  * The lower the number the better.

CONTACTS AND LOCATIONS:
Overall Officials: Lecturer, Study Director — Cairo University
Locations (1):
- CairoU, Cairo, Giza Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No
* The risk that sharing prevents the exploitation of the entire potential of the data obtained.
  * Possible failures in patients' privacy protection.
  * Technical barriers such as the lack of standard formats and possible data misinterpretation.
  * Issues regarding data ownership.
  * Reuse of data for unfair commercial purposes.